CLINICAL TRIAL: NCT04814498
Title: A Phase 1, Open Label, Fixed Sequence Study to Evaluate the Effect of BLD-0409 on the Single Dose Pharmacokinetics of a Cocktail of Probe Substrates for CYP450 Enzymes in Healthy Volunteers
Brief Title: Drug-Drug Interaction (DDI) Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blade Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B-0409-103
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Drug Drug Interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Geneva cocktail (less fexofenadine) & BLD-0409 (Experimental): Following an overnight fast of at least 10 hours, subjects will be administered IP in a fixed sequence.
  Interventions: Drug: Geneva Cocktail; Drug: BLD-0409

INTERVENTIONS:
Drug: Geneva Cocktail — Fixed sequence use of drug cocktail
Drug: BLD-0409 — Fixed sequence use of active product

SUMMARY:
A Phase 1, Open Label, Fixed Sequence Study to Evaluate the Effect of BLD-0409 on the Single Dose Pharmacokinetics of a Cocktail of Probe Substrates for CYP450 Enzymes in Healthy Volunteers

DETAILED DESCRIPTION:
This is a single center, open label study designed to determine the effect of BLD-0409 on the PK of probe substrates and to evaluate the safety and tolerability of BLD-0409 administered alone and co-administered with a cocktail of probe substrates (i.e., Geneva cocktail less fexofenadine) in healthy adult volunteers.

Geneva Cocktail (Less Fexofenadine):

* CYP1A2 Caffeine 50 mg
* CYP2C Flurbiprofen 10 mg
* CYP2C19 Omeprazole 10 mg
* CYP2D6 Dextromethorphan 10 mg
* CYP3A4 Midazolam 1 mg
* CYP2B6 Bupropion 20 mg

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent prior to study entry.
2. Males and females aged 18 to 55 years at the time of consent.
3. Body mass index (BMI) ≥ 18 and ≤ 32 kg/m2.
4. Agree to abstain from alcohol intake from 48 hours before first IP administration through to discharge from the CRU.
5. Agree to abstain from all caffeine- and xanthine-containing products (e.g., coffee, tea, cola drinks, chocolate) for 48 hours before first IP administration through to discharge from the CRU.
6. Have a negative urine drug screen/alcohol breath test at Day -1 (Admission). Repeat urine drug screens will be permitted for suspected false positive results.
7. Use of acceptable contraception.
8. Males must not donate sperm for at least 90 days after the last dose of study drug.
9. Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine or serum pregnancy test on Day -1. If a urine test is conducted and it is positive, a serum pregnancy test must also be performed for confirmation. Females not of childbearing potential must be postmenopausal (defined as cessation of regular menstrual periods for at least 12 months), confirmed by follicle-stimulating hormone (FSH) level > 40 mIU/mL at Screening.
10. In good general health, in the opinion of the Principal Investigator (PI), with no significant medical history, have no clinically significant abnormalities on physical examination at Screening, and/or before administration of the initial dose of study drug.
11. Have clinical laboratory values within normal ranges.

Exclusion Criteria:

1. Active smoker and/or user of nicotine-containing products (i.e., have not used nicotine-containing products within the previous 3 months).
2. Human immunodeficiency virus (HIV) antibody positive.
3. Hepatitis B surface antigen (HBsAg) positive or Hepatitis C virus (HCV) positive.
4. Presence of any underlying or clinically significant physical or psychological medical condition (e.g., hypertension, elevated cholesterol/triglycerides, asthma, or diabetes) that, in the opinion of the PI, would make it unlikely that the subject will complete the study per protocol.
5. History or presence of alcohol or drug abuse (including recreational marijuana use) within the 2 years prior to the first IP administration, and unwillingness to be totally abstinent during the period of confinement.
6. Blood donation or significant blood loss within 30 days prior to the first study drug administration.
7. Plasma donation within 7 days prior to the first study drug administration.
8. Administration of IP in another trial within 30 days prior to the first IP administration, or 5 half-lives, whichever is longer.
9. Females who are pregnant or breastfeeding.
10. Surgery within the past 3 months prior to the first IP administration determined by the PI to be clinically relevant.
11. Consumption of any nutrients known to modulate cytochrome P450 3A4 (CYP3A4) or any strong inhibitors or inducers of CYP3A4, starting from 14 days prior to the first dose of IP on Day 1 and until the EOS assessments.
12. Consumption of cruciferous vegetables or chargrilled meat more than 3 × per week in the previous 2 weeks.
13. Inability to refrain from consumption of grapefruit and Seville oranges or St. John's Wort within 14 days prior to the first dose of IP on Day 1 and until the EOS assessments.
14. Failure to satisfy the PI of fitness to participate for any other reason.
15. Active infection (diagnosed or suspected) or history of recurrent infections.
16. Active malignancy and/or history of malignancy in the past 5 years, except for completely excised non-melanoma skin carcinomas or low grade cervical intraepithelial neoplasia.
17. Serious local infection or systemic infection within 3 months requiring antibiotic treatment.
18. Any acute illness within 30 days prior to Day 1.
19. Use of any prescription or over-the-counter (OTC) medication (except for paracetamol and approved contraceptives) within 5 days or 5 half-lives (whichever is longer) prior to dosing and during course of study without prior approval of the Investigator and Medical Monitor. Simple analgesia (paracetamol) may be permitted at the discretion of the Investigator.
20. For all participants, the use of any estrogen-containing products (e.g., contraceptives, patch, cream, implants) within 14 days prior to the first study drug administration and until the EOS assessments.
21. Inability to refrain from vaccinations within 14 days of the first dose of IP and until the EOS assessments.
22. History of allergy or intolerance to any IP or IP constituents used on study or any clinically significant drug allergy as per the PIs judgment.
23. History of anaphylaxis or other severe allergic reaction to drug, food, toxin, or other exposure.
24. Any surgical or medical condition that could interfere with the absorption, distribution, metabolism, or excretion of the IP.
25. Any evidence of cardiac disease or clinically significant abnormalities on ECG.
26. Systolic blood pressure (BP) > 150 mmHg or < 80 mmHg or diastolic BP > 90 mmHg or < 50 mmHg at Screening with one repeat allowed per the PIs discretion at Screening and Day -1.
27. Heart rate < 40 bpm or > 100 bpm at Screening with one repeat allowed per the PIs discretion at Screening and Day -1.
28. Diets that could alter metabolism (i.e., high protein, Slim Fast®, Nutrisystem®, etc.) within 7 days prior to dosing on Day 1.
29. Weight loss or gain of ≥ 10% in the 30 days prior to dosing.
30. Strenuous exercise, including weightlifting, (> 5 × per week) within 2 weeks prior to first IP administration on Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Area under the drug concentration-time curve from time zero to the last measurable concentration (AUC0-last) | Up to 16 days
  Measured by plasma concentration of probe substrates
Maximum observed drug concentration (Cmax) | Up to 16 days
  Measured by plasma concentration of probe substrates

CONTACTS AND LOCATIONS:
Overall Officials: Kristi McLendon, MD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network Pty Ltd., Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No